CLINICAL TRIAL: NCT06873958
Title: Reducing Postoperative Pneumonia Risk with Spontaneous Breathing Laryngeal Mask Anesthesia in Thoracoscopic Wedge Resection: a Propensity Score Overlap-Weighted Multifactorial Retrospective Cohort Study
Brief Title: Reducing Pneumonia with LMA in Lung Wedge Resection
Status: Not yet recruiting | Type: Observational
Sponsor: Hai Feng (Other)
Responsible Party: Sponsor-Investigator, Hai Feng, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: YXLL-KY-2025(037)
Record Dates: First submitted 2025-03-07; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pneumonia, Postoperative; Anesthesia; Thoracic Surgery; Thoracoscopic Wedge Resection
Keywords: Laryngeal Mask Anesthesia; Spontaneous Breathing; Single-Lung Ventilation; Postoperative Pneumonia; Thoracoscopic Wedge Resection; Propensity Score; Retrospective Cohort Study
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Spontaneous Breathing LMA Group: Patients in this group received general anesthesia using a laryngeal mask airway (LMA) while maintaining spontaneous breathing throughout the procedure. No muscle relaxants were used, and a vagus nerve block was performed to prevent coughing reflexes. Urinary catheters and chest drainage tubes were generally not placed.
- Single-Lung Ventilation Group: Patients in this group received general anesthesia with single-lung isolation and mechanical ventilation. Airway management included double-lumen tubes, single-lumen tubes with bronchial blockers, or LMAs with bronchial blockers. Muscle relaxants were used, and ventilation was controlled.

SUMMARY:
This retrospective cohort study aims to evaluate whether spontaneous breathing laryngeal mask anesthesia (LMA-SBA) reduces the incidence of postoperative pneumonia compared to single-lung isolation mechanical ventilation in patients undergoing thoracoscopic wedge resection. Using propensity score overlap weighting, we will adjust for multiple confounders, including age, COPD, surgical duration, and preoperative laboratory values. Secondary outcomes include postoperative recovery time, fever severity, white blood cell count, neutrophil percentage, length of hospital stay, and ICU admission rate. The study has been approved by the Ethics Committee of the First Affiliated Hospital of Shandong First Medical University (Approval No. YXLL-KY-2025(037)).

DETAILED DESCRIPTION:
Background: Postoperative pneumonia is a significant complication following thoracoscopic wedge resection, potentially linked to the type of anesthesia used. Spontaneous breathing laryngeal mask anesthesia (LMA-SBA) may offer advantages over traditional single-lung isolation mechanical ventilation by preserving natural respiratory function and reducing mechanical ventilation-related lung injury.

Objective: The primary objective is to compare the incidence of postoperative pneumonia between LMA-SBA and single-lung isolation mechanical ventilation groups. Secondary objectives include assessing differences in postoperative recovery time, fever severity, white blood cell count, neutrophil percentage, length of hospital stay, and ICU admission rate.

Methods: This retrospective cohort study will include patients aged ≥18 years who underwent thoracoscopic wedge resection under general anesthesia (LMA-SBA or single-lung isolation mechanical ventilation) at the First Affiliated Hospital of Shandong First Medical University between March 1, 2024, and November 31, 2024. Exclusion criteria include prior thoracic surgery, pleural adhesions, conversion to single-lung isolation during surgery, severe cardiopulmonary dysfunction, and inability to cooperate with postoperative assessments. Data will be collected from electronic medical records, and propensity score overlap weighting will be used to adjust for confounders.

Outcome Measures: Postoperative pneumonia will be diagnosed based on fever (>38°C), cough, new infiltrates on imaging, and abnormal white blood cell count (>10,000/μL or <4,000/μL). Secondary outcomes will be analyzed using weighted regression models.

Ethics: The study protocol has been approved by the Ethics Committee of the First Affiliated Hospital of Shandong First Medical University (Approval No. YXLL-KY-2025(037)).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years ;
2. Patients undergoing thoracoscopic pulmonary wedge resection ;
3. General anesthesia administered intraoperatively (LMA-SBA or endotracheal intubation);
4. Complete preoperative and postoperative clinical data.

Exclusion Criteria:

-

1)History of prior thoracic surgery; 2）Pleural adhesion or pleural effusion caused by tuberculosis or other diseases; 3)Intraoperative conversion from tubeless anesthesia to single-lung isolation-controlled ventilation; 4)Severe cardiopulmonary dysfunction (e.g., history of acute exacerbation of COPD within 1 month preoperatively, patients requiring emergency treatment, or cardiac insufficiency with limited mobility) ; 5)Preoperative neurological dysfunction or sensory abnormalities affecting pain assessment 6)Inability to cooperate with postoperative pain assessment and follow-up 7)Pregnant or breastfeeding women; 8)Patients transferred from other departments with complex comorbidities, prior treatment history, or unstable conditions .

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients undergoing thoracoscopic wedge resection of the lung under general anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2025-03-15 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Incidence of Postoperative Pneumonia | Within 30 days post-surgery
  Postoperative pneumonia is defined based on the American Thoracic Society (ATS) and Infectious Diseases Society of America (IDSA) guidelines, including:
  Fever (body temperature >38°C); Cough, sputum production, or dyspnea; New or progressive infiltrates on chest imaging; Leukocytosis (>10,000/μL) or leukopenia (<4,000/μL). The incidence will be calculated as the proportion of patients diagnosed with pneumonia within 30 days post-surgery.

SECONDARY OUTCOMES:
Postoperative Recovery Time | Immediately after surgery
  Time from the end of anesthesia to the patient's full recovery of consciousness, measured in minutes.
Area Under the Fever Curve Over 3 Days Post-Surgery | First 3 days post-surgery
  The area under the curve (AUC) of body temperature over the first 3 days post-surgery, calculated from temperature measurements taken every 6 hours.
White Blood Cell Count at 24 Hours Post-Surgery | Within 24 hours post-surgery
  White blood cell count measured in peripheral blood within 24 hours after surgery, reported in cells/μL.
Neutrophil Percentage at 24 Hours Post-Surgery | Within 24 hours post-surgery
  Percentage of neutrophils in peripheral blood within 24 hours after surgery.
length of hospital stay after surgery | From surgery to discharge, up to 30 days
  Total number of days from surgery to discharge.
ICU Admission Rate Within 72 Hours Post-Surgery | Within 72 hours post-surgery
  Proportion of patients admitted to the intensive care unit (ICU) within 72 hours after surgery due to any cause.

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong First Medical University, First Affiliated Hospital (Qianfo Mountain Hospital of Shandong Province), Jinan, Shandong, China